CLINICAL TRIAL: NCT05844384
Title: Nanodropper Use in Primary Open-Angle Glaucoma Patients: A Non-Inferiority Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: 59th Medical Wing (U.S. Federal Agency)
Collaborators: Nanodropper, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: C.2022.041
Record Dates: First submitted 2023-02-14; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Ocular Hypertension; Primary Open Angle Glaucoma
Keywords: Nanodropper; Primary Open Angle Glaucoma; Microdrops; Ocular Hypertension
MeSH Terms: conditions — Ocular Hypertension; Glaucoma, Open-Angle

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, single-masked, active-controlled, crossover (AB:BA)
Who Masked: Investigator
Masking Description: The investigators performing the vision assessment and measuring the intraocular pressure are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Nanodroper (Experimental): * Patients are given a Nanodropper to use with their IOP-lowering eyedrops.
  * Patient returns for a safety check 1 month following the start of Nanodropper use.
  * At 3 months, the patient returns for clinical assessment and starts using IOP-lowering eyedrops without Nanodropper for 3 months.
  * The patient returns at 6 months for final clinical assessment
  Interventions: Device: Nanodropper
- Regular Dropper (Active Comparator): * Patient continues using current IOP-lowering eyedrops without Nanodropper adaptor.
  * At 3 months, the patient returns for clinical assessment and starts using IOP-lowering eyedrops with Nanodropper for 3 months.
  * Patient returns for a safety check 1 month following the start of Nanodropper use.
  * The patient returns at 6 months for final clinical assessment
  Interventions: Device: Regular dropper

INTERVENTIONS:
Device: Nanodropper — Nanodropper delivers 1/5 of eye drop volume compared to regular droppers
  Arms: Nanodroper
Device: Regular dropper — Delivers full eye drop volume
  Arms: Regular Dropper

SUMMARY:
This randomized, single-masked, crossover, non-inferiority trial aims to evaluate the safety and efficacy of Nanodropper-mediated microdrops of ocular hypotensive topical treatments (experimental intervention) compared to standard drops of the same medication(s) (active comparator) in Wilford Hall Ambulatory Surgical Center (WHASC) primary open-angle glaucoma (POAG) and ocular hypertension (OHTN) patients.

DETAILED DESCRIPTION:
The primary objective of this study is to compare changes in intraocular pressure (IOP) in a population of POAG and OHTN patients in response to administration of 1) standard drops of IOP lowering medications and 2) Nanodropper-mediated microdrops of IOP-lowering medications. The hypothesis is that Nanodropper-mediated microdrops of IOP-lowering medications will not result in a significant difference in IOP relative to standard drops of IOP-lowering medications after three months of daily eyedrop administration with each delivery system. The primary outcome measure for this efficacy endpoint will be mean IOP (mm Hg) ± SEM. A secondary objective of this trial is to evaluate Nanodropper's safety and usability. Surveys that have been designed to gain an understanding of the differences in side effects and usability between using Nanodropper-mediated microdrops compared to standard eyedrops will be administered to patients at the enrollment visit and at each follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* POAG/OHTN patients above the age of 18 years.
* On a maximum of 2 IOP lowering medications.
* Stable disease without progression in IOP, optic disc cupping, RNFL changes, and visual field changes within the previous 1 year.

Exclusion Criteria:

* Glaucoma not of the POAG or OHTN variety or other retinal diseases.
* Progression of disease within the preceding 1 year (IOP elevation, optic disc cupping, visual field changes).
* Using more than 2 IOP-lowering medications.
* IOP-lowering surgical interventions or lasers except for SLT. SLT may have been completed 6+ months prior to study start date.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-17 (Actual); Primary Completion 2024-03-17 (Estimated); Study Completion 2024-03-17 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in mean intraocular pressure at 6 month | Change from baseline to month 6
  Change in mean intraocular pressure (unit = mmHg) from baseline to month 6 measure with applanation tonometer

SECONDARY OUTCOMES:
Change from baseline in mean high contrast visual acuity at 6-month | Change from baseline to month 6
  Change in the mean uncorrected visual acuity (unit = logMAR) from baseline to month 6 measure with ETDRS chart from baseline at 6 months post-op.
Change from baseline in mean retinal nerve fiber layer thickness at 6-month | Change from baseline to month 6
  Change in the mean retinal nerve fiber layer thickness (unit = micrometer) from baseline to month 6 measure with optical coherence tomographer.
Change from baseline in visual field mean deviation at 6-month | Change from baseline to month 6
  Change in the visual field mean deviation (unit = decibels) from baseline to month 6measure with Humphreys Visual Field Analyzer.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Papp, MD, Principal Investigator — 59th Medical Wing
Locations (1):
- Wilford Hall Ambulatory Surgical Center, Lackland Air Force Base, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Result of the study will be published in a scientific journal upon completion.

DOCUMENTS (1):
  • Informed Consent Form (2022-03-17): https://cdn.clinicaltrials.gov/large-docs/84/NCT05844384/ICF_000.pdf